CLINICAL TRIAL: NCT04087200
Title: The Protective Effect of Early High Dose High-intensity Statins on Cardiovascular and Renal Events in Patients With Acute Coronary Syndrome
Brief Title: Protective Effect of Early High Dose stATins On Cardiovascular and Renal Events in Acute Coronary Syndrome
Acronym: PRATO-ACS
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiopatici Toscani (Other)
Collaborators: Azienda USL 4 Prato (Other)
Responsible Party: Principal Investigator, Anna Toso, Principal Investigator, Centro Cardiopatici Toscani
Other Study IDs: OSS 15.161
Record Dates: First submitted 2019-08-30; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Acute Coronary Syndrome
Keywords: STEMI; NSTEMI; Acute kidney injury; Renal function; Statin therapy
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Registration of all ACS patients (STEMI and NSTEMI) admitted to the cardiology ward and scheduled for early invasive strategy. The aim is to evaluate the protective effects of early (on admission) high-dose high-potency statin therapy on early and mid-term cardiac and renal events in this subset of patients.

DETAILED DESCRIPTION:
Statin-naive patients and those on statin therapy with ACS who are admitted to the cardiology ward of our public (National Health Service) hospital and are scheduled for early invasive strategy receive immediately on admission, always before angiographic procedure, high-dose statin therapy. Either atorvastatin 80 mg or rosuvastatin 40 mg is administered at the discretion of the physician. During hospitalization various pertinent cardiac and renal parameters, including hematological, angiographic, clinical data are registered in a dedicated database. Clinical follow-up and hematological analysis are done 1 month after discharge. A second follow-up, either clinical or by telephone, is done 1 year after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome (ST elevation and non ST elevation)
* Early invasive strategy

Exclusion Criteria:

* contraindication to statin therapy
* refusal of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Statin-naive patients and those on statin therapy with ACS (both STEMI and NSTEMI)
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute renal function changes | Within 72 hours after hospital admission
  Changes in creatinine and/or cystatine values
Inflammatory profile changes | up to 1 month
  Changes from baseline in CRP values
Lipid profile changes | up to 1 month
  Changes from baseline in cholesterol values
Platelet count | up to 1 month
  Changes from baseline in platelet count
Platelet volume | up to 1 month
  Changes from baseline in platelet volume
Platelet aggregation profile | up to 1 month
  Changes from baseline in platelet reactivity (Verify Now)

SECONDARY OUTCOMES:
Major cardiovascular adverse events | up to 12 months
  Death, myocardial infarction, stroke or coronary revascularization
Renal function changes | Changes from baseline at 1 month
  glomerular filtration rate
Major adverse cardiovascular and renal adverse events | up to 1 month
  Death, myocardial infarction, stroke, coronary revascularization or glomerular filtration rate reduction > = 25% compared to baseline

OTHER OUTCOMES:
Impact of age and frailty profile on primary and secondary outcomes | Up to 1 month
  Frailty evaluation (combination of FRAIL scale questionnaire and hand-grip strength measurement)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Division, Prato Hospital, Prato, Italy